Official Title: Prevalence of Chronic Inebriates to the Emergency Department and Suitability for Sobering

**House Services** 

NCT #: NCT01783223

Date: March 13, 2011

## **Project Summary Study proposal**

This study is intended to evaluate the prevalence of chronically inebriated patients in the Emergeny Department (ED). Patients will be identified prospectively by screening all patients (24/7) presenting to the ED for one month. A running tally of all patients in the ED will be kept. Of these patients, any patient that is noted to have alcohol intoxication will be identified. The chart of that patient will be reviewed for details about the patient's alcohol use and for the patient's suitability for a sobering house, which is a place where intoxicated patients can go to await sobriety. The chart will also be reviewed for the number of previous visits for alcohol use to our hospital ever and in the last year.

This study is a prospective cross sectional study investigating the prevalence of intoxicated patients presenting to the Emergency Department and the number who can be discharged to a sobering center. All patients presenting to the ED will be screened. Patients who screen positive for alcohol intoxication (patient reported complaint, provider diagnosis, or positive ethanol measurement) will be enrolled in this sub study. Patients under 18, prisoners, and pregnant patients will be excluded.

## Background

It has been extensively documented that a small number of emergency department patients make disproportionate use of the emergency department. These users tend to be poor, homeless, socially isolated, have alcohol and drug problems, and lack insurance (Stern et al 1991, Baker et al 1994). These patterns have prompted extensive investigation into alcohol abuse and the role of the emergency department.

While all these studies have shown improved outcomes with each respective intervention, the problem of length of intervention and specific determinants for effectiveness are raised. Few studies have looked at particular patterns within subgroups of problematic drinkers. Kelly et al investigated the consumption patterns, alcohol related problems and predictors of problematic drinking among adolescents who visit the ER. The authors were able to identify three pieces of information available in the initial assessment, which would identify them as problem drinkers, and may require further intervention.

No studies however have been able to accurately depict the inebriate population that is responsible for so many ED visits annually, as well as the number of EMS runs annually (70% of those who use EMS >5 times annually are intoxicated patients (Brokaw et al 1998)). This small group of ED patients accounts for a large percentage of the visits and costs of services provided in emergency departments. Definitions of heavy use in the literature vary ,though a majority of studies that focus specifically on this group and setting use a definition of four or more visits per 12-15 months (Malone 1995).

The recommendations from the 2002 conference "Alcohol Problems among Emergency Department Patients: Research on Identification and Intervention" include investigating how cultural and demographic factors affect patients' access to services for alcohol-related problems, delivery of those services in ED's, and patient outcomes (Hungerford 2002). A method of decreasing the use of Emergency Department's by intoxicated individual's that has been proposed is to instead observe intoxicated patients in sobering centers that would provide observation for transfer to a higher level of care for patients with medical emergencies, and could provide a suitable environment for intervention. The number of patients that may benefit from this level of care is not known The goal of this study was to determine how many patients that are seen in the Emergency Department with alcohol intoxication as part or all of their care, and how many would be able to be seen in a sobering center rather than the ED if it were available.

## Study Design

Observational cohort

This is a prospective observational study of all patients presenting to the ED of an urban, Level 1 trauma centers. All patients arriving to the ED will be screened prospectively by trained research associates 24 hours a day and seven days a week during the study period in one month increments. Patients with a presenting complaint of alcohol intoxication or who are diagnosed with alcohol intoxication will be included

When an intoxicated patient is identified, study information will be collected. This will include patient demographics, diagnoses, vital signs including heart rate, blood pressure, oxygen saturation and respiratory rate, blood alcohol concentration (BAC), GCS on arrival, ability to ambulate independently on arrival, use of physical or chemical restraint, previous ED visits, length of stay, disposition, the suitability of the patient for transfer to a sobering center, and health insurance will be collected. Suitability for transfer to a sobering center is at the discretion of the treating physician and includes the ability to ambulate without assistance.

Data will be stored without identifying information. Data will be analyzed using descriptive statistics

**Anticipated Benefit(s) to Study Participants** 

None.

**Potential Risks to Study Participants** 

None.